CLINICAL TRIAL: NCT05324098
Title: Leveraging Technology (STAND-T) to Achieve Equity for Men With Prostate Cancer on Androgen Deprivation Therapy
Brief Title: Leveraging Technology to Achieve Equity for Men With Prostate Cancer on Androgen Deprivation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Myovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 215514; NCI-2022-02225 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: Health Technologies
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health services research (STAND-T, text messages) (Experimental): Patients review educational material and resources via online STAND-T platform. Patients also receive interactive text messages for 3 months.
  Interventions: Other: STAND-T platform; Other: Survey Administration; Other: Text Messages

INTERVENTIONS:
Other: STAND-T platform — Internet-based intervention comprised of evidence-based, patient materials and resources
  Other Names: STAND-T
Other: Survey Administration — Satisfaction and follow-up surveys will be administered to participants
Other: Text Messages — Participants will receive periodic text messages
  Other Names: Short Message Service (SMS) Text

SUMMARY:
This clinical trial studies a digital platform, the supportive therapy in androgen deprivation (STAND-T), in achieving equity for men undergoing treatment with androgen deprivation therapy for prostate cancer. STAND-T is a digital platform that provides prostate health information, evidence-based materials and resources. STAND-T may help improve health, address symptoms, and promote equity in men with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess study feasibility of the STAND-T program at the Helen Diller Family Comprehensive Cancer Center (HDFCCC) and Zuckerberg San Francisco General Hospital and Trauma Center (ZSFG) genitourinary (GU) medical, surgical, and radiation oncology practices.

SECONDARY OBJECTIVE:

I. To measure preliminary estimates of acceptability and usage of a digital platform, STAND-T.

EXPLORATORY OBJECTIVE:

I. To describe diet (e.g., fruit and vegetable intake), lifestyle (e.g., moderate to vigorous exercise, smoking status), clinical (symptoms e.g., fatigue), and health related quality of life (QoL) outcomes (e.g., sleep disturbance), physiologic measures (body mass index, BMI) at baseline and change in these metrics from baseline to 3 months post-intervention.

OUTLINE:

Patients review educational material and resources via online STAND-T platform. Patients also receive interactive text messages for 3 months.

After completion of study, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Ability to understand study procedures and to comply with them for the entire length of the study
* Ability of individual or legal guardian/representative to understand an informed consent document and the willingness to sign it
* Adenocarcinoma of the prostate
* Current or planned anti-androgen therapy (ADT) (oral or injection) with gonadotropin-releasing hormone (GnRH) antagonist or luteinizing hormone releasing hormone (LHRH) agonist
* Life expectancy duration of 6 months or longer from date of study consent
* Prior and concurrent radiation is allowed
* Treatment with concurrent androgen signaling inhibitors is allowed
* < 75 minutes/week of vigorous aerobic exercise based on Godin survey or < 2 days per week of vigorous activity

Exclusion Criteria:

* Contraindication to any study-related procedure or assessment
* Planned surgery/chemotherapy/immunotherapy/parp inhibitor treatment during the study period
* Prior and concurrent investigational therapies
* Unable to read/speak English
* Unable to access the Internet
* Has seen an exercise counselor in the past 6 months for prostate or cardiovascular health
* Has seen a dietary counselor in the past 6 months for prostate or cardiovascular health

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Completion rate | Up to 3 months
  The point estimation and 95% confidence interval (CI) of the percentage of participants who complete the 3-month study will be obtained overall and by race/ethnicity and geography.

SECONDARY OUTCOMES:
Participants reported satisfaction level | Up to 3 months
  Satisfaction will be measured on a likert scale: Extremely Unsatisfied, Dissatisfied, Neither Satisfied or Dissatisfied, Satisfied, Extremely Satisfied. The point estimation and 95% CI of the percentage (95% CI) of participants who are satisfied or extremely satisfied with the program at 3 months will be obtained.
Change in the proportion of men who were Extremely Satisfied/Satisfied | Up to 3 months
  Satisfaction will be measured on a likert scale: Extremely Unsatisfied, Dissatisfied, Neither Satisfied or Dissatisfied, Satisfied, Extremely Satisfied. Change in the percentage (proportion) of men who were Extremely Satisfied/Satisfied from 7 days to 3 months will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Kenfield, DSc, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang EY, Borno HT, Washington Iii SL, Friedlander T, Zhang S, Trejo E, Van Blarigan EL, Chan JM, Shariff-Marco S, Beatty AL, Kenfield SA. Engaging Men of Diverse Racial and Ethnic Groups With Advanced Prostate Cancer in the Design of an mHealth Diet and Exercise Intervention: Focus Group Study. JMIR Cancer. 2023 Jun 1;9:e45432. doi: 10.2196/45432. PMID 37261885